CLINICAL TRIAL: NCT06802497
Title: Comparison of Early Postoperative Outcomes of Patients Undergoing Laparoscopic Lateral Suspension and V-NOTES Lateral Suspension With the Salman Ketenci Gencer Technique
Brief Title: Comparison of Postoperative Outcomes of Laparoscopic Lateral Suspension and V-NOTES Lateral Suspension With the Salman Ketenci Gencer Technique
Status: Recruiting | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: GaziosmanpasaTREHfkg
Record Dates: First submitted 2025-01-04; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: laparoscopy; v-notes lateral suspension; pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients underwent laparoscopic lateral suspension
- patients underwent V-NOTES lateral suspension with SalmanKetenciGencer technique

SUMMARY:
Comparison of Early Postoperative Outcomes of Patients Undergoing Laparoscopic Lateral Suspension and V-NOTES Lateral Suspension with the Salman Ketenci Gencer Technique

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 3 or 4 pelvic organ prolapse Sexually active patients

Exclusion Criteria:

* Cervical pathology History of loop electrosurgical excision procedure (LEEP) or conization Presence of vaginal, pelvic, or adnexal mass Suspicious abdominal malignancy Morbid obesity Any pelvic infection Signs of pregnancy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study planned to include 84 patients with pelvic organ prolapse.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Improvement in Pelvic Organ Prolapse (POP) Severity by POP-Q Score | 6 months
  POP-Q measurements assess the degree of pelvic organ prolapse in patients, using a combined system that includes multiple parameters to evaluate the anterior and posterior vaginal walls, cervix, and vaginal vault. This study will compare the POP-Q values of patients following laparoscopic lateral suspension and V-Notes lateral suspension with the Salmanketencigencer technique to assess improvements in prolapse severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)